CLINICAL TRIAL: NCT04458298
Title: A Two-Stage, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of OP-101 (Dendrimer N-acetyl-cysteine) in Patients With Severe COVID-19
Brief Title: A Study to Evaluate OP-101 (Dendrimer N-acetyl-cysteine) in Severe Coronavirus Disease 2019 (COVID-19) Patients
Acronym: PRANA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Ashvattha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: OP-101-004
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: SARS-COV-2; Coronavirus; Cytokine storm; Acute respiratory distress syndrome; Inflammation; IL-6; Treatment; OP-101
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Cytokine Release Syndrome; Respiratory Distress Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Stage I: Cohort A: OP-101 2 mg/kg (Experimental): Participants will receive a single intravenous (IV) infusion of OP-101 2 milligram per kilogram (mg/kg) on Day 1.
  Interventions: Drug: OP-101
- Stage I: Cohort B: OP-101 4 mg/kg (Experimental): Participants will receive a single IV infusion of OP-101 4 mg/kg on Day 1.
  Interventions: Drug: OP-101
- Stage I: Cohort C: OP-101 8 mg/kg (Experimental): Participants will receive a single IV infusion of OP-101 8 mg/kg on Day 1.
  Interventions: Drug: OP-101
- Stage I: Cohort D: Placebo (Placebo Comparator): Participants will receive a single IV infusion of matching placebo on Day 1.
  Interventions: Drug: Placebo
- Stage II: Cohort E: OP-101 8 mg/kg (Experimental): Participants will receive a single IV infusion of OP-101 8 mg/kg on Days 1 and 4.
  Interventions: Drug: OP-101
- Stage II: Cohort F: Placebo (Placebo Comparator): Participants will receive a single IV infusion of matching placebo on Days 1 and 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OP-101 — OP-101 infusion will be administered intravenously.
  Arms: Stage I: Cohort A: OP-101 2 mg/kg; Stage I: Cohort B: OP-101 4 mg/kg; Stage I: Cohort C: OP-101 8 mg/kg; Stage II: Cohort E: OP-101 8 mg/kg
Drug: Placebo — Matching placebo infusion will be administered intravenously.
  Arms: Stage I: Cohort D: Placebo; Stage II: Cohort F: Placebo

SUMMARY:
The primary purpose of Stage-I of this study is to evaluate the safety and tolerability of OP-101 in patients with severe COVID-19 and of Stage 2 of this study is to evaluate the efficacy of OP-101 in patients with severe COVID-19.

The secondary purpose of Stage 1 and Stage 2 of this study is to determine the effect of OP-101 reducing proinflammatory cytokines biomarkers in severe COVID-19 Patients.

A further secondary objective of Stage 2 of this study is:

To evaluate the safety and tolerability of OP-101 in patients with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Stage I:

* Body mass index (BMI) less than or equal to (<=) 35 kilogram per meter square (kg/m^2)
* Positive laboratory test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or respiratory infection with recent exposure to a person with laboratory-proven SARS-CoV-2
* Patient has an ordinal scale score between 5 and 7, inclusive, using the WHO 7OS
* Hypoxemia defined by saturation of peripheral oxygen (SpO2) of less than (<) 95 percent (%) on room air or Acute respiratory distress syndrome (ARDS)
* Occurrence of at least two of the following criteria: fever greater than (>) 38.0 degree celsius, tachycardia >90 beats/minute, tachypnea >20 breaths/minute, leucocytosis >12*109 per liter (/L) or leucopoenia <4 *10^9/L
* Enrollment must occur within 72 hours from the initiation of mechanical ventilation or high-flow oxygen
* A signed informed consent form (ICF) from the patient or the patient's legally authorized representative must be available (telephone consent is acceptable)
* Female patients may not be pregnant, lactating, or breastfeeding
* Female patients of childbearing potential must have negative result for pregnancy test at screening
* Male patients must agree to use a barrier method of contraception during the study and for 90 days after the last dose
* Participants must have an estimated glomerular filtration rate of greater than or equal to (>=) 45 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) at screening
* Must agree not to enroll in another study of an investigational agent prior to completion of this study.

Stage II:

* Positive laboratory test for SARS-CoV-2 or respiratory infection with recent exposure to a person with laboratory-proven SARS-CoV-2
* Patient has an ordinal scale score between 5 and 8, inclusive, using the WHO 10OS.
* Patients with an ordinal score of 5 must be receiving oxygen by mask at a rate of 10 L or greater
* Hypoxemia defined by SpO2 of <95% on room air or diagnosed with ARDS
* Hyperinflammation (elevated CRP > upper limit of local normal for laboratory range) at screening
* A signed ICF from the patient or the patient's legally authorized representative must be available (telephone consent is acceptable)
* Female patients may not be pregnant, lactating, or breastfeeding
* Female patients of childbearing potential must have negative result for pregnancy test at screening
* Patients must have an estimated glomerular filtration rate of >= 30 mL/min/1.73 m^2 at screening
* Male patients must agree to use a barrier method of contraception during the study and for 90 days after the last dose
* Must agree not to enroll in another study of an investigational agent prior to completion of this study.

Exclusion Criteria:

Stage I:

* Not expected to survive for more than 24 hours
* Underlying clinical condition where, in the opinion of the investigator, it would be extremely unlikely that the patient would come off ventilation (eg, motor neuron disease, Duchenne muscular dystrophy, or rapidly progressive interstitial pulmonary fibrosis)
* Severe chronic obstructive pulmonary disease requiring long-term home oxygen therapy or mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure used solely for sleep-disordered breathing
* Congestive heart failure, defined as New York Heart Association Class IV
* Acute left ventricular failure or myocardial infarction
* Currently receiving extracorporeal membrane oxygenation (ECMO) therapy
* Receiving renal dialysis therapy for chronic renal failure
* Moderate to severe liver failure (Childs-Pugh Score >12)
* Presence of any active malignancy (other than nonmelanoma skin cancer) that required treatment within the last 2 years
* Lung transplant patient
* WHO Class III or IV pulmonary hypertension
* Documented deep venous thrombosis or pulmonary embolism within past 3 months
* Major trauma in the preceding 5 days
* Concurrent treatment with immune modulatory study drugs (e.g., anti-IL6 antibodies, Janus kinase (JAK) kinase inhibitors) or other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 within 30 days or 5 half-lives, whichever is longer, prior to dosing with OP-101; except for those that have received FDA emergency-use authorization and have become standard of care (SOC). Concurrent treatment with corticosteroids is permitted if participant has documented continued hypoxemia (SpO2 of <95% on room air) and hyper-inflammation (CRP>=10 mg/L) at screening.
* Has lost or donated >450 mL of whole blood or blood products within 30 days before screening
* Has any finding that, in the view of the investigator or medical monitor, would compromise the patient's safety requirements
* Is employed by the Sponsor, the contract research organization, or the study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, contract research organization, or study site employee.

Stage II:

* Not expected to survive for more than 24 hours
* Underlying clinical condition where, in the opinion of the investigator, it would be extremely unlikely that the patient would come off ventilation (e.g., motor neuron disease, Duchenne muscular dystrophy, or rapidly progressive interstitial pulmonary fibrosis)
* Severe chronic obstructive pulmonary disease requiring long-term home oxygen therapy or mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure used solely for sleep-disordered breathing
* Congestive heart failure, defined as New York Heart Association Class IV
* Acute left ventricular failure or myocardial infarction
* Currently receiving ECMO therapy
* Receiving renal dialysis therapy for end stage renal disease
* Moderate to severe liver failure (Childs-Pugh Score >12)
* Presence of any active malignancy (other than nonmelanoma skin cancer) that required treatment within the last 2 years
* Lung transplant patient
* WHO Class III or IV pulmonary hypertension
* Documented deep venous thrombosis or pulmonary embolism within past 3 months
* Major trauma in the preceding 5 days
* Concurrent treatment with approved or emergency use authorized immune modulatory study drugs (eg, anti-IL6 antibodies [tocilizumab], JAK kinase inhibitors [baricitinib]) or other investigational agents with actual or possible direct acting antiviral activity against SARS-CoV-2 within 30 days or 5 half-lives, whichever is longer, before dosing with OP-101.
* Has lost or donated >450 mL of whole blood or blood products within 30 days before screening
* Mechanical ventilation for >72 hours at the time of dosing
* Has any finding that, in the view of the investigator or medical monitor, would compromise the patient's safety requirements
* Is employed by the Sponsor, the contract research organization, or the study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, contract research organization, or study site employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Stage I: Number of Participants with Treatment Emergent Adverse Events Graded as Assessed by CTCAE Version 4.0 | Up to Day 60
  Number of participants with treatment emergent adverse events will be evaluated as a measure of safety and tolerability of OP-101 by monitoring and documenting all adverse events, which include laboratory test variables.
Stage II: Percentage of Participants Who Were Alive (i.e., not died due to any reason) at Day 29 | Day 29

SECONDARY OUTCOMES:
Stage I: Time to Improvement (2 points) in Clinical Status Assessment Using the World Health Organization 7-Point Ordinal Scale (WHO 7OS) | Up to Day 30
  WHO-7 is a 7 point ordinal scale for clinical improvement with scores ranging from 0 to 7 where 0= uninfected, 1= no limitation of activities (ambulatory), 2= limitation of activities (ambulatory), 3= hospitalized, no oxygen therapy (hospitalized mild disease), 4= Hospitalized, oxygen by mask or nasal prongs (hospitalized mild disease), 5= Hospitalized, noninvasive ventilation or high-flow oxygen (hospitalized severe disease), 6= Hospitalized, intubation and mechanical ventilation (hospitalized severe disease), 7= Hospitalized, ventilation + additional organ support - pressors, renal replacement therapy, ECMO.
Stage I: Time to Resolution of Fever for at least 48 hours Without Antipyretics for Patients with Documented Fever (>=37.2 degree celsius [oral], or >=37.8 degree celsius [rectal], or >=38.0 degree celsius [tympanic]) | Up to Day 30
Stage I: Time to Improvement in Oxygenation for at least 48 hours | Up to Day 30
  Improvement in oxygenation is defined by increase in pulse oxygen saturation/fraction of inspired oxygen (SpO2/FiO2) of >=50 compared with nadir SpO2/FiO2.
Stage I: Change from Baseline in the World Health Organization (WHO)-7 Point Ordinal Scale | Baseline up to Day 30
  WHO-7 is a 7 point ordinal scale for clinical improvement with scores ranging from 0 to 7 where 0= uninfected, 1= no limitation of activities (ambulatory), 2= limitation of activities (ambulatory), 3= hospitalized, no oxygen therapy (hospitalized mild disease), 4= Hospitalized, oxygen by mask or nasal prongs (hospitalized mild disease), 5= Hospitalized, noninvasive ventilation or high-flow oxygen (hospitalized severe disease), 6= Hospitalized, intubation and mechanical ventilation (hospitalized severe disease), 7= Hospitalized, ventilation + additional organ support - pressors, renal replacement therapy, ECMO.
Stage I: Time to Discharge from Clinic or Hospital or to National Early Warning Score 2 (NEWS2) of <=2 and maintained for 24 hours | Up to Day 30
  NEWS2 consists of: Physiological Parameters: Respiration rate (per minute), SpO2 Scale 1 (%), SpO2 Scale 2 (%), Use of Air or oxygen, Systolic blood pressure (mmHg), Pulse (per minute), Consciousness, Temperature (°C).
Stage I: Percentage of Patients Alive and not Using Supplemental Oxygen at Time of Discharge from Hospital/Clinic or Day 30 | Up to Day 30
Stage I: Number of Days of Resting Respiratory Rate of more than 24 breath/min | Up to Day 30
Stage I: Number of Days with Hypoxemia | Up to Day 30
  Hypoxemia is defined by Saturation of Peripheral Oxygen (SpO2) of less than (<) 95 percent (%) on room air or acute respiratory distress syndrome (ARDS).
Stage I: Number of Days of Supplemental Oxygen use | Up to Day 30
Stage I: Number of Ventilator-free Days | Up to Day 28
Stage I: Number of Days in Intensive Care Unit (ICU) | Up to Day 30
Stage I: Number of Days of Hospitalization for Survivors | Up to Day 30
Stage I: Number of Participants with all cause Deaths | Up to Day 30
Stage I: Percent Change from Baseline in Proinflammatory Cytokines | Baseline up to Day 30
  Percent change from baseline in proinflammatory cytokines (C-reactive protein [CRP], ferritin, and interleukin-6 [IL-6]) will be reported.
Stage I: Incidence of Drug-related Serious Adverse Events (SAEs) | Up to Day 60
Stage II: Percentage of Participants Who Were Alive and free of Respiratory Failure | Up to Day 29
  Respiratory failure is defined as at least 1 of the following: i. Endotracheal intubation and mechanical ventilation; ii. Oxygen delivered by high-flow nasal cannula (>20 L/minute; >=50% oxygen) OR fraction of inspired oxygen >50% delivered by Face Mask, Venturi, Rebreather Mask, Oxymizer Mask; iii. Non-invasive positive pressure oxygen - Continuous Positive Airway Pressure (CPAP) use for chronic sleep apnea treatment is not included in the definition of respiratory failure; iv. Extracorporeal membrane oxygenation (ECMO).
Stage II: Percentage of Participants Alive and Free of Invasive Mechanical Ventilation | Up to Day 29
Stage II: Percentage of Participants Alive and Discharged From the Hospital | Up to Day 29
Stage II: Percentage of Participants Alive and not Using Supplemental Oxygen at Time of Discharge from Hospital/Clinic or Day 29 | Up to Day 29
Stage II: Percent Change from Baseline in Proinflammatory Biomarkers | Baseline up to Day 29
  Percent change from baseline in proinflammatory cytokines (CRP, ferritin, IL-6, and serum neurofilament light chain [sNfL]) will be reported.
Stage II: Number of Days in Intensive Care Unit (ICU) | Up to Day 29

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, Loma Linda, California
  - Research site, Fort Lauderdale, Florida
  - Research site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research site, Baltimore, Maryland
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Amarillo, Texas
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No